CLINICAL TRIAL: NCT00055874
Title: Treatment Optimization Trial in Chronic Myeloid Leukemia (CML) - Randomized Controlled Comparison of Imatinib vs. Imatinib/Interferon-alpha vs. Imatinib/Low-Dose AraC vs. Interferon-alpha Standard Therapy and Determination of the Role of Allografting in Newly Diagnosed Chronic Phase
Brief Title: Imatinib Mesylate With or Without Interferon Alfa or Cytarabine Compared With Interferon Alfa Followed by Donor Stem Cell Transplant in Treating Patients With Newly Diagnosed Chronic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. h.c. R. Hehlmann, Investigator, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: III-MK-CML-IV; CDR0000271424 (Registry Identifier: PDQ (Physician Data Query)); EU-20248
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2011-11

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Interferon-alpha; Cytarabine; Hydroxyurea; Imatinib Mesylate; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: cytarabine
Drug: hydroxyurea
Drug: imatinib mesylate
Procedure: allogeneic bone marrow transplantation
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy before a donor bone marrow transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. Also, imatinib mesylate may stop the growth of cancer cells by blocking the enzymes needed for cancer cell growth. Interferon alfa may interfere with the growth of cancer cells and slow the growth of cancer. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. It is not yet known which treatment regimen is most effective in treating chronic phase chronic myelogenous leukemia.

PURPOSE: This randomized phase III trial is studying imatinib mesylate with or without interferon alfa or cytarabine to see how well it works compared with interferon alfa followed by donor stem cell transplant in treating patients with newly diagnosed chronic phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the hematologic, cytogenetic, and molecular response rates in patients with newly diagnosed chronic phase chronic myelogenous leukemia treated with imatinib mesylate alone or with interferon alfa or low-dose cytarabine vs interferon alfa standard therapy.
* Compare the group-dependent, progression-free and overall survival and time to progression in patients treated with these regimens.
* Compare the efficacy of allogeneic stem cell transplantation vs imatinib mesylate-based therapy in patients eligible for transplantation.
* Compare the efficacy of reduced-intensity conditioning vs standard conditioning in patients over 45 years of age.
* Determine the time to and duration of hematologic, cytogenetic, and molecular responses and correlate these factors in patients treated with these regimens.
* Compare the short- and long-term adverse effects of these regimens in these patients.
* Compare the presentation, duration, and responses to therapy of accelerated and blastic phases in patients treated with these regimens.
* Determine the survival of high-risk patients after early allografting.
* Determine the influence of pre-transplantation therapies on the outcome of allogeneic stem cell transplantation in these patients.

OUTLINE: This is a randomized, multicenter, pilot study. Patients are stratified according to participating center. Patients with low- to intermediate-risk disease are randomized to 1 of 4 treatment arms. Patients with high-risk disease are randomized to 1 of 3 treatment arms with imatinib mesylate-based regimens.

* Arm I: Patients receive oral imatinib mesylate once daily for up to 12 months in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral imatinib mesylate as in arm I. Patients also receive interferon alfa subcutaneously (SC) 3 times a week beginning at least 3 months after the start of imatinib mesylate.
* Arm III: Patients receive oral imatinib mesylate as in arm I. Patients also receive cytarabine SC up to twice daily for 5 days monthly beginning at least 3 months after the start of imatinib mesylate.
* Arm IV: After initial cytoreduction with hydroxyurea, patients receive interferon alfa SC daily with or without hydroxyurea. In the absence of a complete response after 3 months, patients may also receive low-dose cytarabine SC once daily. Treatment continues for up to 21 months.

Patients who fail interferon alfa therapy are crossed over to receive imatinib mesylate.

Patients who fail therapy with imatinib mesylate and are eligible for an allogeneic transplantation are stratified according to availability of donor (HLA-identical related vs unrelated), status, and participating center. Patients are randomized to receive an allogeneic transplantation or continue any salvage therapy.

Patients who are not eligible for allogeneic transplantation receive hydroxyurea and cytarabine or high-dose chemotherapy with autologous stem cell rescue followed by interferon- or imatinib mesylate-based therapy.

Patients over 45 years of age are further randomized to receive an age-adjusted standard conditioning regimen or reduced intensity preparative regimen (mini transplantation) prior to allogeneic transplantation.

Patients are followed every 6 months for 3 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,600 patients (400 per treatment arm) will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed chronic phase chronic myelogenous leukemia (CML)

  * bcr-abl positive
  * No blasts, promyelocytes, myelocytes, or metamyelocytes in the peripheral blood
* Availability of a HLA-identical sibling or unrelated donor

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No second malignancy requiring therapy
* No evidence of disease-related symptoms or extramedullary disease (including hepatosplenomegaly)
* No serious diseases that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior interferon

Chemotherapy

* No prior chemotherapy other than hydroxyurea

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* Not specified

Other

* Prior anagrelide allowed
* No participation in another clinical trial

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1551 (Actual)
Dates: Start 2002-06; Primary Completion 2012-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Overall survival
Risk group-dependent survival
Progression-free survival
Hematologic, cytogenetic, and molecular response rates

SECONDARY OUTCOMES:
Adverse drug effects
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ruediger Hehlmann, MD, Study Chair — III. Medizinische Klinik Mannheim
Locations (66):
- Germany (65):
  - Krankenhaus / Klinikum Krefeld, Aachen
  - Kreiskrankenhaus Aurich, Aurich
  - Kreiskrankenhaus, Bad Hersfeld
  - St. Hedwig Krankenhaus, Berlin
  - Haematologisch-Onkologische Schwerpunktpraxis, Berlin
  - Schwerpunktpraxis fuer Haematologie und Internistische Onkologie, Berlin
  - Gemeinschaftspraxis fuer Haematologie und Internistische Onkologie, Berlin
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld
  - Augustinum, Bonn
  - Hamatologische Sprechstunde, Brandenburg
  - Praxis Dres. F.& G. Doering, Bremen
  - Staedtisches Kliniken Delmenhorst, Delmenhorst
  - Universitaetsklinikum Essen, Essen
  - Evangelisches Krankenhaus Essen Werden, Essen
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Internistische Praxisgemeinschaft, Germering
  - DR Herbert - Nieper Krankenhaus Goslar, Goslar
  - Universitaetsklinikum Goettingen, Göttingen
  - St. Marien Hospital - Katholisches Krankenhaus Hagen gGmbH, Hagen
  - Asklepios Klinik St. Georg, Hamburg
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Evangelische Krankenhaus Hamm, Hamm
  - Medizinische Universitaetsklinik und Poliklinik, Heidelberg
  - Universitatsklinikum Heidelberg, Heidelberg
  - Ruprecht - Karls - Universitaet Heidelberg, Heidelberg
  - Medical University Hospital Homburg, Homburg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - St. Vincentius - Kliniken, Karlsruhe
  - Klinikum Kempten Oberallgaeu, Kempten
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Klinikum Krefeld GmbH, Krefeld
  - Internistisches Fachaerzte Zentrum Langen, Langen
  - Caritas - Krakenhaus Lebach, Lebach
  - Onkologische Schwerpunktpraxis - Leer, Leer
  - Klinikum Lippe - Lemgo, Lemgo
  - Klinikum der Stadt Ludwigshafen am Rhein, Ludwigshafen am Rhein
  - III Medizinische Klinik Mannheim, Mannheim
  - Hospital Maria-Hilf II, Mönchengladbach
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Haematologische Schwerpunktpraxis, Munich
  - Krankenhaus Muenchen Schwabing, München
  - Haematologisch - Onkologische Gemeinschaftspraxis - Muenster, Münster
  - Hematologische Onkologische Praxis, Regensburg
  - Klinikum der Universitaet Regensburg, Regensburg
  - Klinikum Remscheid GmbH, Remscheid
  - Internistische Schwerpunktpraxis, Rüsselsheim am Main
  - Diakonie - Krankenhaus, Schwäbisch Hall
  - St. Marien - Krankenhaus Siegen GMBH, Siegen
  - Kreiskrankenhaus Siegen, Siegen
  - Hanse-Klinikum Stralsund - Krankenhaus West, Stralsund
  - Onkologische Schwerpunktpraxis - Straubing, Straubing
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Haematologische Praxis, Stuttgart
  - Klinik fuer Onkologie - Katharinenhospital Stuttgart, Stuttgart
  - Diakonie Klinikum Stuttgart, Stuttgart
  - Trier
  - Schwerpunktpraxis fuer Rheumatologie und Haematologie/Internistische Onkologie, Tübingen
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
  - Haematologische Praxis, Weiden
  - Praxis Fuer Haemotologie Und Internistischer Onkologie, Wuppertal
  - Helios Kliniken Wuppertal University Hospital, Wuppertal
  - Hamatologisch - Onkologische Praxis Wurzburg, Würzburg
  - University Wurzburg, Würzburg
- Basel, Switzerland

REFERENCES:
- [Result] Hehlmann R, Lauseker M, Jung-Munkwitz S, Leitner A, Muller MC, Pletsch N, Proetel U, Haferlach C, Schlegelberger B, Balleisen L, Hanel M, Pfirrmann M, Krause SW, Nerl C, Pralle H, Gratwohl A, Hossfeld DK, Hasford J, Hochhaus A, Saussele S. Tolerability-adapted imatinib 800 mg/d versus 400 mg/d versus 400 mg/d plus interferon-alpha in newly diagnosed chronic myeloid leukemia. J Clin Oncol. 2011 Apr 20;29(12):1634-42. doi: 10.1200/JCO.2010.32.0598. Epub 2011 Mar 21. PMID 21422420
- [Result] Burchert A, Muller MC, Kostrewa P, Erben P, Bostel T, Liebler S, Hehlmann R, Neubauer A, Hochhaus A. Sustained molecular response with interferon alfa maintenance after induction therapy with imatinib plus interferon alfa in patients with chronic myeloid leukemia. J Clin Oncol. 2010 Mar 10;28(8):1429-35. doi: 10.1200/JCO.2009.25.5075. Epub 2010 Feb 8. PMID 20142590
- [Result] Saussele S, Lauseker M, Gratwohl A, Beelen DW, Bunjes D, Schwerdtfeger R, Kolb HJ, Ho AD, Falge C, Holler E, Schlimok G, Zander AR, Arnold R, Kanz L, Dengler R, Haferlach C, Schlegelberger B, Pfirrmann M, Muller MC, Schnittger S, Leitner A, Pletsch N, Hochhaus A, Hasford J, Hehlmann R; German CML Study Group. Allogeneic hematopoietic stem cell transplantation (allo SCT) for chronic myeloid leukemia in the imatinib era: evaluation of its impact within a subgroup of the randomized German CML Study IV. Blood. 2010 Mar 11;115(10):1880-5. doi: 10.1182/blood-2009-08-237115. Epub 2009 Nov 18. PMID 19965667
- [Derived] Saussele S, Hehlmann R, Fabarius A, Jeromin S, Proetel U, Rinaldetti S, Kohlbrenner K, Einsele H, Falge C, Kanz L, Neubauer A, Kneba M, Stegelmann F, Pfreundschuh M, Waller CF, Oppliger Leibundgut E, Heim D, Krause SW, Hofmann WK, Hasford J, Pfirrmann M, Muller MC, Hochhaus A, Lauseker M. Defining therapy goals for major molecular remission in chronic myeloid leukemia: results of the randomized CML Study IV. Leukemia. 2018 May;32(5):1222-1228. doi: 10.1038/s41375-018-0055-7. Epub 2018 Feb 26. PMID 29479070
- [Derived] Saussele S, Krauss MP, Hehlmann R, Lauseker M, Proetel U, Kalmanti L, Hanfstein B, Fabarius A, Kraemer D, Berdel WE, Bentz M, Staib P, de Wit M, Wernli M, Zettl F, Hebart HF, Hahn M, Heymanns J, Schmidt-Wolf I, Schmitz N, Eckart MJ, Gassmann W, Bartholomaus A, Pezzutto A, Leibundgut EO, Heim D, Krause SW, Burchert A, Hofmann WK, Hasford J, Hochhaus A, Pfirrmann M, Muller MC; Schweizerische Arbeitsgemeinschaft fur Klinische Krebsforschung and the German CML Study Group. Impact of comorbidities on overall survival in patients with chronic myeloid leukemia: results of the randomized CML study IV. Blood. 2015 Jul 2;126(1):42-9. doi: 10.1182/blood-2015-01-617993. Epub 2015 Apr 27. PMID 25918346
- [Derived] Lauseker M, Hasford J, Hoffmann VS, Muller MC, Hehlmann R, Pfirrmann M; German CML Study Group. A multi-state model approach for prediction in chronic myeloid leukaemia. Ann Hematol. 2015 Jun;94(6):919-27. doi: 10.1007/s00277-014-2246-2. Epub 2014 Dec 3. PMID 25465231
- [Derived] Hanfstein B, Lauseker M, Hehlmann R, Saussele S, Erben P, Dietz C, Fabarius A, Proetel U, Schnittger S, Haferlach C, Krause SW, Schubert J, Einsele H, Hanel M, Dengler J, Falge C, Kanz L, Neubauer A, Kneba M, Stegelmann F, Pfreundschuh M, Waller CF, Spiekermann K, Baerlocher GM, Pfirrmann M, Hasford J, Hofmann WK, Hochhaus A, Muller MC; SAKK and the German CML Study Group. Distinct characteristics of e13a2 versus e14a2 BCR-ABL1 driven chronic myeloid leukemia under first-line therapy with imatinib. Haematologica. 2014 Sep;99(9):1441-7. doi: 10.3324/haematol.2013.096537. Epub 2014 May 16. PMID 24837466
- [Derived] Proetel U, Pletsch N, Lauseker M, Muller MC, Hanfstein B, Krause SW, Kalmanti L, Schreiber A, Heim D, Baerlocher GM, Hofmann WK, Lange E, Einsele H, Wernli M, Kremers S, Schlag R, Muller L, Hanel M, Link H, Hertenstein B, Pfirrman M, Hochhaus A, Hasford J, Hehlmann R, Saussele S; German Chronic Myeloid Leukemia Study Group; Schweizerische Arbeitsgemeinschaft fur Klinische Krebsforschung (SAKK). Older patients with chronic myeloid leukemia (>/=65 years) profit more from higher imatinib doses than younger patients: a subanalysis of the randomized CML-Study IV. Ann Hematol. 2014 Jul;93(7):1167-76. doi: 10.1007/s00277-014-2041-0. PMID 24658964
- [Derived] Lauseker M, Hasford J, Pfirrmann M, Hehlmann R; German CML Study Group. The impact of health care settings on survival time of patients with chronic myeloid leukemia. Blood. 2014 Apr 17;123(16):2494-6. doi: 10.1182/blood-2013-11-539742. Epub 2014 Mar 12. PMID 24622328
- [Derived] Hehlmann R, Muller MC, Lauseker M, Hanfstein B, Fabarius A, Schreiber A, Proetel U, Pletsch N, Pfirrmann M, Haferlach C, Schnittger S, Einsele H, Dengler J, Falge C, Kanz L, Neubauer A, Kneba M, Stegelmann F, Pfreundschuh M, Waller CF, Spiekermann K, Baerlocher GM, Ehninger G, Heim D, Heimpel H, Nerl C, Krause SW, Hossfeld DK, Kolb HJ, Hasford J, Saussele S, Hochhaus A. Deep molecular response is reached by the majority of patients treated with imatinib, predicts survival, and is achieved more quickly by optimized high-dose imatinib: results from the randomized CML-study IV. J Clin Oncol. 2014 Feb 10;32(5):415-23. doi: 10.1200/JCO.2013.49.9020. Epub 2013 Dec 2. PMID 24297946
- [Derived] Kalmanti L, Saussele S, Lauseker M, Proetel U, Muller MC, Hanfstein B, Schreiber A, Fabarius A, Pfirrmann M, Schnittger S, Dengler J, Falge C, Kanz L, Neubauer A, Stegelmann F, Pfreundschuh M, Waller CF, Spiekermann K, Krause SW, Heim D, Nerl C, Hossfeld DK, Kolb HJ, Hochhaus A, Hasford J, Hehlmann R; German Chronic Myeloid Leukemia Study Group; Schweizerische Arbeitsgemeinschaft fur Klinische Krebsforschung (SAKK). Younger patients with chronic myeloid leukemia do well in spite of poor prognostic indicators: results from the randomized CML study IV. Ann Hematol. 2014 Jan;93(1):71-80. doi: 10.1007/s00277-013-1937-4. Epub 2013 Oct 27. PMID 24162333